CLINICAL TRIAL: NCT05377424
Title: Acute Adenosine Receptor Antagonism to Promote Breathing Plasticity in ALS
Brief Title: Adenosine 2A Receptor Antagonism and AIH in ALS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: ALS Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB202101568; OCR41682 (Other: UF OnCore)
Record Dates: First submitted 2022-04-26; First posted 2022-05-17 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: ALS
Keywords: ALS; hypoxia; breathing; istradefylline
MeSH Terms: conditions — Hypoxia; Respiratory Aspiration | interventions — istradefylline; Insemination, Artificial, Homologous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AIH + istradefylline (AIH+IST) (Experimental): Participants enrolled in this study arm will ingest a 20mg tablet containing istradefylline. Four hours later, participants will receive acute intermittent hypoxia (AIH). Breathing and pinch strength will be tested prior to taking the medication, and then immediately before, 60 minutes and 120 minutes after AIH. Participants will breathe 15 episodes/session of acute low oxygen. Air concentrations will be monitored to ensure delivery of 1-minute episodes of low oxygen, with 2 minutes room-air intervals. Respiratory rate, oxygen saturation, heart rate/rhythm, and blood pressure will be monitored throughout the session.
  Interventions: Drug: Consume 20mg of istradefylline; Other: Low Oxygen therapy
- Sham-AIH + istradefylline (sham+IST) (Active Comparator): This is a sham counterpart to the low oxygen. Participants enrolled in this study arm will ingest a 20mg tablet containing istradefylline. Four hours later, participants will receive SHAM acute intermittent hypoxia (SHAM). Breathing and pinch strength will be tested prior to taking the medication, and then immediately before, 60 minutes and 120 minutes after SHAM. Participants will breathe 15 episodes/session of sham low oxygen, in which normal air is used. One-minute episodes of sham low oxygen are separated by 2 minutes room-air intervals. Respiratory rate, oxygen saturation, heart rate/rhythm, and blood pressure will be monitored throughout the session.
  Interventions: Drug: Consume 20mg of istradefylline; Other: SHAM counterpart to low oxygen therapy.
- AIH + placebo (AIH+CON) (Active Comparator): This is a placebo counterpart to the istradefylline drug. Participants enrolled in this study arm will ingest a 20mg tablet containing microcrystalline cellulose. Four hours later, participants will receive acute intermittent hypoxia (AIH). Breathing and pinch strength will be tested prior to taking the medication, and then immediately before, 60 minutes and 120 minutes after AIH. Participants will breathe 15 episodes/session of acute low oxygen. Air concentrations will be monitored to ensure delivery of 1-minute episodes of low oxygen, with 2 minutes room-air intervals. Respiratory rate, oxygen saturation, heart rate/rhythm, and blood pressure will be monitored throughout the session.
  Interventions: Other: Low Oxygen therapy; Drug: Placebo counterpart to the istradefylline drug
- Sham-AIH + placebo (sham+CON) (Active Comparator): This is a sham counterpart to low oxygen, and a placebo counterpart to the istradefylline drug. Participants enrolled in this study arm will ingest a 20mg tablet containing microcrystalline cellulose. Four hours later, participants will receive SHAM acute intermittent hypoxia (SHAM). Breathing and pinch strength will be tested prior to taking the medication, and then immediately before, 60 minutes and 120 minutes after SHAM. Participants will breathe 15 episodes/session of sham low oxygen, in which normal air is used. One-minute episodes of sham low oxygen are separated by 2 minutes room-air intervals. Respiratory rate, oxygen saturation, heart rate/rhythm, and blood pressure will be monitored throughout the session.
  Interventions: Drug: Placebo counterpart to the istradefylline drug; Other: SHAM counterpart to low oxygen therapy.

INTERVENTIONS:
Drug: Consume 20mg of istradefylline — Consume a single 20 mg istradefylline tablet
  Other Names: Nourianz
  Arms: AIH + istradefylline (AIH+IST); Sham-AIH + istradefylline (sham+IST)
Other: Low Oxygen therapy — Breathing short periods of low oxygen, consisting of 15 episodes of 1 minute of breathing 10% oxygen, with 2 minutes of breathing 21% oxygen. 45 minutes total.
  Other Names: Acute Intermittent Hypoxia; AIH
  Arms: AIH + istradefylline (AIH+IST); AIH + placebo (AIH+CON)
Drug: Placebo counterpart to the istradefylline drug — Consume a single microcrystalline cellulose
  Other Names: Placebo
  Arms: AIH + placebo (AIH+CON); Sham-AIH + placebo (sham+CON)
Other: SHAM counterpart to low oxygen therapy. — Breathing short periods of sham low oxygen, consisting of 15 episodes of 1 minute of breathing 21% oxygen, separated by 2 minutes of breathing 21% oxygen. 45 minutes total.
  Other Names: SHAM acute intermittent hypoxia; SHAM-AIH
  Arms: Sham-AIH + istradefylline (sham+IST); Sham-AIH + placebo (sham+CON)

SUMMARY:
The purpose of this research study is to determine the effects of a medication, istradefylline, in conjunction with breathing air with reduced oxygen for short periods of time (called acute intermittent hypoxia, or AIH), on breathing. This project will study breathing in people with amyotrophic lateral sclerosis (ALS) and unaffected, age-matched adults. Istradefylline is prescribed to increase movement in people with other neuromuscular conditions. A recently completed study found that people with ALS took deeper breaths, 60 minutes after using AIH.

DETAILED DESCRIPTION:
This repeated measures, placebo-controlled, randomized study will study feasibility and efficacy of istradefylline, an adenosine 2A receptor antagonist in conjunction with acute intermittent hypoxia (AIH).

Participation in this study includes a screening for eligibility, plus 4 individual study visits separated by 1 week. The eligibility screening will include a review of medical history and medications, along with a breathing test and sleep study.

Each participant will experience a different study condition on each of their 4 study visits: an "AIH + istradefylline" (AIH+IST) visit, and a "sham-AIH + istradefylline" (sham+IST) visit, an "AIH + placebo (AIH+CON)" visit, and a "sham-AIH + placebo" (sham+CON) visit. The visits will be in random order for each subject. Participants and the testing investigators will not be told which order the visits will be. Participants need to avoid exercise and caffeine and nicotine products for >8 hours before each study visit.

AIH + istradefylline visit: participants will take 20 mg of istradefylline. After a 4-hour break, participants will receive a 45-minute session of AIH, consisting of 15, one-minute periods of low oxygen (10% O2) with two-minute periods of normal oxygen (21% O2).

Sham AIH + istradefylline visit: participants will take 20 mg of istradefylline. After a 4-hour break, participants will receive a 45-minute session of SHAM AIH, consisting of 15, one-minute intervals of normal oxygen (21% O2) with two-minute periods of normal oxygen (21% O2).

AIH + placebo visit: participants will take 20 mg of microcrystalline cellulose. After a 4-hour break, participants will receive a 45-minute session of AIH, consisting of 15, one-minute periods of low oxygen (10% O2) with two-minute periods of normal oxygen (21% O2).

Sham AIH + placebo visit: participants will take 20 mg of microcrystalline cellulose. After a 4-hour break, participants will receive a 45-minute session of SHAM AIH, consisting of 15, one-minute intervals of normal oxygen (21% O2) with two-minute periods of normal oxygen (21% O2).

Venous blood samples will be collected at the start of each visit as general safety labs (complete blood count, uric acid, blood chemistry), and to assess levels of istradefylline levels in the blood. Additional blood tests 4 and 6 hours later will measure changes in serum istradefylline.

The study will assess vital signs, patient-reported symptoms, resting breathing, strength of the breathing muscles, and maximal voluntary pinch force at the start of each visit. These measures will then be repeated 1 and 2 hours after AIH or SHAM. Throughout the AIH and SHAM interventions, respiratory rate, oxygen saturation, end-tidal carbon dioxide (CO2), heart rate, and blood pressure will be monitored.

For the primary efficacy endpoint, the study will measure breath volume at the start of each visit, and 1 and 2 hours after the AIH and SHAM interventions. A linear mixed model will be used to compare differences in tidal volume. Main effects include treatment and time, with participants as random effects.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking adults aged 21-80 years will be eligible to participate.

   - Upon screening, eligible patients will have an
2. ALS diagnosis (El Escorial diagnostic classifications of probable/definite ALS),
3. vital capacity (VC) > 60% of predicted value, and
4. ALS Functional Rating Scale (ALSFRS-R) scores of 2 or greater for bulbar and respiratory items: swallowing, speech, salivation, dyspnea, orthopnea, and respiratory insufficiency.
5. Additionally, patients taking riluzole and/or edaravone must be on a stable dose for >30 days.
6. Unaffected control subjects will be eligible if they have a vital capacity (VC) > 60% of predicted value.

Exclusion Criteria:

Patient and control are ineligible if they

1. are pregnant
2. have an active respiratory infection,
3. took antibiotics within 4 weeks,
4. are diagnosed with another neurodegenerative disease,
5. have symptomatic cardiovascular disease or dysrhythmias (resting tachycardia and hypertension),
6. exhibit history or presence of hypoxemia or hypercapnia,
7. presence of rest tachypnea (RR ˃30),
8. have a BMI >35 kg/m2,
9. have a seizure disorder,
10. take respiratory inhalers daily for airway disease, or
11. require external respiratory support while awake and upright, or
12. supplemental oxygen at rest or at night.
13. In addition, the following conditions are exclusionary for the use of istradefylline: routine use of CYP3A4 inducers (i.e. carbamazepine, phenobarbitol, rifampin, phenytoin, St. John's Wort, glucocorticoids) or
14. medications that may suppress ventilation, history of moderate renal impairment or severe hepatic impairment, and history of hallucinations or psychosis.
15. Patients who cannot safety swallow thin liquids (required for administration of istradefylline and placebo) will also be ineligible.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Treatment differences in the rate of adverse events. | Through study completion (an average of 4-6 weeks)
  Any reported adverse events will be tracked and recorded.
Change in resting tidal volume | 120 minutes after AIH
  Averaged volume of breaths at rest

SECONDARY OUTCOMES:
Serum Istradefylline | 4 hours post- istradefylline or placebo
  Blood test to measure change in level of istradefylline
Serum Istradefylline | 6 hours post- istradefylline or placebo
  Blood test to measure change in level of istradefylline
Subject-reported involuntary movements | 4 hours post- istradefylline or placebo
  Participants will use a 0-10 scale to report the intensity of any involuntary movements or tremors. (a higher number would correspond to more involuntary movements or tremors)
Change in minute ventilation | 120 minutes post-intervention.
  Change in the average volume of air during a minute of resting breathing.

OTHER OUTCOMES:
Change in maximal voluntary pinch force | 120 minutes post-intervention.
  Pinch force of the thumb will be evaluated in a seated position.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Smith, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Clinical and Translational Research Building, Gainesville, Florida
  - UF Health Jacksonville, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trumbower RD, Jayaraman A, Mitchell GS, Rymer WZ. Exposure to acute intermittent hypoxia augments somatic motor function in humans with incomplete spinal cord injury. Neurorehabil Neural Repair. 2012 Feb;26(2):163-72. doi: 10.1177/1545968311412055. Epub 2011 Aug 5. PMID 21821826
- [Background] Vivodtzev I, Tan AQ, Hermann M, Jayaraman A, Stahl V, Rymer WZ, Mitchell GS, Hayes HB, Trumbower RD. Mild to Moderate Sleep Apnea Is Linked to Hypoxia-induced Motor Recovery after Spinal Cord Injury. Am J Respir Crit Care Med. 2020 Sep 15;202(6):887-890. doi: 10.1164/rccm.202002-0245LE. No abstract available. PMID 32369393
- [Background] Seven YB, Simon AK, Sajjadi E, Zwick A, Satriotomo I, Mitchell GS. Adenosine 2A receptor inhibition protects phrenic motor neurons from cell death induced by protein synthesis inhibition. Exp Neurol. 2020 Jan;323:113067. doi: 10.1016/j.expneurol.2019.113067. Epub 2019 Oct 17. PMID 31629857
- [Background] Sajjadi E, Seven YB, Ehrbar JG, Wymer JP, Mitchell GS, Smith BK. Acute intermittent hypoxia and respiratory muscle recruitment in people with amyotrophic lateral sclerosis: A preliminary study. Exp Neurol. 2022 Jan;347:113890. doi: 10.1016/j.expneurol.2021.113890. Epub 2021 Oct 6. PMID 34624328
- [Derived] Sales de Campos P, Smith-Hublou M, Olsen WL, Souza Leite W, Wymer JP, Napoli NJ, Vose AK, Pulley MT, Mitchell GS, Smith BK. Acute Adenosine Receptor Antagonism in Combination With Acute Intermittent Hypoxia to Promote Breathing Plasticity in Amyotrophic Lateral Sclerosis: Protocol for a Randomized, Double-Blinded, Placebo-Controlled Trial. JMIR Res Protoc. 2025 Nov 7;14:e76105. doi: 10.2196/76105. PMID 41202295